CLINICAL TRIAL: NCT03861117
Title: Impact of the Combination of Pressure Support and Positive End Expiratory Pressure During Spontaneous Breathing Trial Versus T-piece on the Time to Successful Extubation
Brief Title: Pressure Support and Positive End Expiratory Pressure During Spontaneous Breathing Trial
Acronym: SBT-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0982; 2019-A00106-51 (Other: ID-RCB)
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Critically Ill Adult Patients With Difficult Weaning
Keywords: Critical care; spontaneous breathing trial; T-piece; positive end-expiratory pressure; difficult weaning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assisted strategy (Experimental): Ability to be weaned is determined with pressure support and positive end-expiratory pressure.
  Interventions: Procedure: Assisted strategy
- Non assisted strategy (Active Comparator): Ability to be weaned is determined with T-piece.
  Interventions: Procedure: Non assisted strategy

INTERVENTIONS:
Procedure: Assisted strategy — Daily spontaneous breathing trial (SBT) with 7 cmH2O pressure support and 5 cmH2O positive end-expiratory pressure are performed to assess weanability. In case of success, a SBT with T-piece is performed to determine if the patients is at high risk of extubation failure. In this case and/or in the presence of risk factors, systematic non-invasive ventilation is applied after extubation.
  Arms: Assisted strategy
Procedure: Non assisted strategy — Daily spontaneous breathing trials (SBT) with T-piece are performed to assess weanability. In the presence of risk factors, systematic non-invasive ventilation is applied after extubation.
  Arms: Non assisted strategy

SUMMARY:
The aim of this study is to assess if a bundle associating pressure support and positive end-expiratory pressure during spontaneous breathing trial and detection by T-piece of patients with high-risk of extubation failure can reduce the time to successful extubation in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years old or more
* Intubated and ventilated in intensive care unit for more than 24 hours
* Patient ready for weaning evaluation
* Failure of a first T-piece SBT

Exclusion Criteria:

* Chronic neuromuscular disease
* Guillain-Barré Syndrome
* Central nervous system disease with consciousness disorder
* Tracheostomy
* Chronic disease with life expectancy less than 1 year
* Pregnancy, breast feeding
* Withholding life support regarding a reintubation
* Prisoner or patient interned in psychiatric hospital
* Guardianship
* Language barrier
* Lack of medical insurance
* Lack of the patient's consent (or of the next of kin where appropriate)
* Patient under an exclusion period after enrollment in another research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Time (hours) to successful extubation | 90 days
  Successful extubation is defined as extubation without retintubation within the 7 following days.

SECONDARY OUTCOMES:
Rate of first extubation | 90 days
  percentage (%) of patients with a first successful extubation divided by the total number of patients per group
Invasive mechanical ventilation duration | 90 days
  time (hours) spent on invasive mechanical ventilation since inclusion
duration of non-invasive and invasive mechanical ventilation | 90 days
  time (hours) spent on invasive or non mechanical ventilation since inclusion
ventilator-free days at Day 90 | 90 days
  90 minus the number of days spent on invasive mechanical ventilation (days) since inclusion. Zero day is allocated to dead patients.
Intensive care unit length of stay | 90 days
  time (days) spent in intensive care unit from inclusion until discharge or death
hospital length of stay | 90 days
  time (days) spent in the hospital from inclusion until discharge or death
Day 90 mortality | 90 days
  percentage (%) of patients dead at Day 90
reintubation rate | 90 days
  percentage (%) of the number of patients with any reintubation divided by the number of patients per group

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix-Rousse, Lyon, France

REFERENCES:
- [Background] Mezidi M, Yonis H, Chauvelot L, Danjou W, Dhelft F, Bazzani A, Girard M, Bitker L, Richard JC. Pressure support and positive end-expiratory pressure versus T-piece during spontaneous breathing trial in difficult weaning from mechanical ventilation: study protocol for the SBT-ICU study. Trials. 2022 Dec 12;23(1):993. doi: 10.1186/s13063-022-06896-4. PMID 36503500
- [Result] Mezidi M, Yonis H, Chauvelot L, Deniel G, Dhelft F, Gaillet M, Noirot I, Folliet L, Chabert P, David G, Danjou W, Baboi L, Bettinger C, Bernon P, Girard M, Provoost J, Bazzani A, Bitker L, Richard JC. Spontaneous breathing trial with pressure support on positive end-expiratory pressure and extensive use of non-invasive ventilation versus T-piece in difficult-to-wean patients from mechanical ventilation: a randomized controlled trial. Ann Intensive Care. 2024 Apr 17;14(1):59. doi: 10.1186/s13613-024-01290-6. PMID 38630372